## STATISTICAL ANALYSIS PLAN

## TITLE: Evaluation of Vitamin D With And Without Hormonal Contraception on Sexual Function in Women With Polycystic Ovary Syndrome

**INVESTIGATORS:** Steven R. Lindheim, MD, MMM; Lisa Kellar, MD; Logan Havermann, Michelle Durrant, MD; Rose Maxwell, PhD

October 14, 2016

NCT02865187

Statistical analysis will consist of 1) comparison of baseline with 6 month scores on FSFI total and subscale scores, and comparison of baseline with 6 month Vitamin D levels. Paired t-test will be used to determine degree of change and statistical significance of change scores.